CLINICAL TRIAL: NCT00469599
Title: Treatment of Secondary Hyperparathyroidism in the Uremic Patient. A Study Comparing Alfacalcidol and Paricalcitol
Brief Title: Treatment of Secondary Hyperparathyroidism in the Uremic Patient
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated after 86 pt included, because of recruitment problems
Sponsor: Zealand University Hospital (Other)
Responsible Party: Ditte Hansen MD, Roskilde County Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2006-005981-37
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-04

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease; Vitamin D Deficiency
Keywords: Hyperparathyroidism, Secondary; Kidney Failure, Chronic; Renal Insufficiency, Chronic; Vitamin D Deficiency; Renal Osteodystrophy; Hemodialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Vitamin D Deficiency; Kidney Failure, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — paricalcitol; alfacalcidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): alfacalcidol 16 weeks, 6 weeks wash out, paricalcitol 16 weeks
  Interventions: Drug: paricalcitol
- 2 (Active Comparator): paricalcitol ´16 weeks, 6 weeks wash out, alfacalcidol 16 weeks
  Interventions: Drug: alfacalcidol

INTERVENTIONS:
Drug: paricalcitol — 3 microg 3 times a week. dosage is increased/decreased 50 % every second week according to iPTH, ionised s-calcium and phosphate
  Other Names: Zemplar
  Arms: 1
Drug: alfacalcidol — 1 microg 3 times a week, dosage is titrated every second week according to iPTH, phosphate and ionised s-calcium.
  Arms: 2

SUMMARY:
The purpose of this study is to compare alfacalcidol and paricalcitol in the treatment of secondary hyperparathyroidism in hemodialysis patients.

DETAILED DESCRIPTION:
Secondary hyperparathyroidism is a common feature in patients with chronic kidney disease. Its clinical consequences include renal osteodystrophy, calciphylaxia and potentially vascular calcifications with increased morbidity and mortality.

Reduced synthesis of active vitamin D contributes to secondary hyperparathyroidism. Therefore we primarily manage this condition with activated vitamin D. In Denmark alfacalcidol is the primary choice of vitamin D analog.

However hypercalcemia and hyperphosphatemia may limit the use of alfacalcidol therapy due to increased risk of vascular calcification and mortality.

Therefore a new vitamin D analog, paricalcitol, has been developed, that may be less prone to develop hypercalcemia and hyperphosphatemia.

However a randomised controlled clinical study comparing alfacalcidol and paricalcitol has never been performed.

The primary objective of this study is to evaluate the effect of alfacalcidol and paricalcitol on intact parathyroid hormone level and the tendency towards hyperphosphatemia and hypercalcemia.

The study is performed in 117 patients with end stage renal failure on maintenance hemodialysis therapy in 6 different Danish hemodialysis units.

The design is a multicenter crossover study where patients are randomized into two treatment arms. After a wash out period of 6 weeks they are receiving alfacalcidol or paricalcitol for a period of 16 weeks and after a further wash out period of 6 weeks they receive the contrary treatment (respectively paricalcitol or alfacalcidol) for 16 weeks.

The initial dose of alfacalcidol (1 μg intravenously after dialysis) and paricalcitol (3 μg intravenously after dialysis) will be adjusted every second week based on iPTH, p-calcium and p-phosphate.

P-calcium, p-phosphate, iPTH, pulse and blood pressure are measured every second week. By the beginning and the end of each period of treatment, alkaline phosphatase, 25OH-D3, 1,25 (OH)2 vitamin D and safety parameters are measured, pulse wave velocity and pulse wave analysis is performed in a subgroup.

Alfacalcidol and paricalcitol are both registered treatment modalities for patients with renal failure and secondary hyperparathyroidism and should not perform any risk for the safety of the enrolled patients as well as the blood sampling and blood pressure measurement should not perform any risk either.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. Secondary hyperparathyroidism; iPTH > 350 pg/ml before any treatment or after 6 weeks without any treatment with vitamin D.
3. Chronic renal insufficiency receiving hemodialysis.
4. P-phosphate < 1,8 mmol/l
5. P-calcium ion < 1,25 mmol/l
6. Receiving maximal possible dose of calcium-based phosphate binder.
7. Accepting 2 x 6 weeks without vitamin D.
8. Safe anti conception in fertile women
9. Do not expect need of calcimimetics or parathyroidectomy during the next year.
10. Written informed consent.

Exclusion Criteria:

1. Malignancy
2. Disease or condition making the patient unable to participate
3. Expected lifetime less than one year.
4. Pregnancy and nursing
5. Allergic to contents of Zemplar or Etalpha
6. Currently receiving calcimimetics
7. Participating in other clinical intervention studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-07; Primary Completion 2010-09 (Estimated); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The effect of alfacalcidol and paricalcitol on intact parathyroid hormone level and the tendency towards hyperphosphatemia and hypercalcemia | 16 weeks

SECONDARY OUTCOMES:
alkaline phosphatase, 25OH-vitamin D,1,25 OH2-vitamin D,calcium x phosphate product, blood pressure, pulse, pulse pressure, parathyroidectomy, pulse wave velocity and pulse wave analysis, initiation of treatment with calcimimetics. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ditte Hansen, MD, Principal Investigator — Zealand University Hospital
Locations (8):
- Denmark (8):
  - Holbæk County Hospital, Holbæk, Holbæk
  - Holstebro County Hospital, Holstebro, Holstebro
  - Roskilde County Hospital, Roskilde, Roskilde
  - Aalborg University Hospital, Aalborg
  - Århus University Hospital Skejby, Aarhus
  - Hospital of Southwest Denmark Esbjerg, Esbjerg
  - Odense University Hospital, Odense
  - Viborg County Hospital, Viborg

REFERENCES:
- [Derived] Hansen D, Rasmussen K, Rasmussen LM, Bruunsgaard H, Brandi L. The influence of vitamin D analogs on calcification modulators, N-terminal pro-B-type natriuretic peptide and inflammatory markers in hemodialysis patients: a randomized crossover study. BMC Nephrol. 2014 Aug 12;15:130. doi: 10.1186/1471-2369-15-130. PMID 25112372
- [Derived] Hansen D, Brandi L, Rasmussen K. Treatment of secondary hyperparathyroidism in haemodialysis patients: a randomised clinical trial comparing paricalcitol and alfacalcidol. BMC Nephrol. 2009 Sep 24;10:28. doi: 10.1186/1471-2369-10-28. PMID 19778452